CLINICAL TRIAL: NCT03458481
Title: A Multicenter, Randomized, Parallel Assigned, Open-label Study to Investigate the Efficacy and Safety of Yimitasvir Phosphate (DAG181)/Sofosbuvir(SOF) Combination for 12 Weeks in Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Phase 2 Study of Yimitasvir Phosphate Capsules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DDAG181PA-16-005
Record Dates: First submitted 2018-02-10; First posted 2018-03-08 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Chronic HCV Infection
Keywords: Chronic Genotype 1 HCV Infection
MeSH Terms: interventions — Sofosbuvir; yimitasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOF+DAG181 100 mg (Experimental): Patients with genotype 1 HCV infection without cirrhosis will receive SOF+DAG181 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: DAG181
- SOF+DAG181 200 mg (Experimental): Patients with genotype 1 HCV infection without cirrhosis will receive SOF+DAG181 200 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: DAG181

INTERVENTIONS:
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: sofosbuvir; Sovaldi®
Drug: DAG181 — Capsule administered orally once daily
  Other Names: Yimitasvir

SUMMARY:
The safety, tolerability and antiviral activity of DAG181/SOF in treatment-naive and treatment-experienced patients with chronic hepatitis C virus (HCV) genotype 1 infection

DETAILED DESCRIPTION:
A phase 2, multicenter, randomized, parallel Assigned, open-label study to explore the safety, tolerability and antiviral activity of DAG181/SOF combination for 12 weeks in adult subjects with chronic genotype 1 HCV infection.

Approximately 120 HCV genotype 1 subjects without cirrhosis will be enrolled, treatment-experienced subjects are ≤20%, all subjects will be randomized (1:1) to one of the following two treatment groups by IWRS (Medidata Balance): a) DAG181 100 mg/ SOF 400 mg once daily for 12 weeks, b) DAG181 200 mg/ SOF 400 mg once daily for 12 weeks. Randomization will be stratified by "treatment-naive" or "treatment-experienced".

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Male or female, age≥18 years;
3. A female subject is eligible to enter the study if it is confirmed that she is:

   1. Of non-childbearing potential (i.e., women who have had a hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal-women > 50 years of age with cessation (for≥12 months) of previously occurring menses), or
   2. Of childbearing potential (Women≤50 years of age with amenorrhea will be considered to be of childbearing potential). These women must have a negative serum pregnancy test at screening, and must use specific contraceptive methods from screening until 4 weeks after last dose of study drugs, such as complete abstinence from intercourse, vaginal ring, cervical cap or contraceptive diaphragm, IUD, etc.
4. All male study subjects must agree to consistently and correctly use specific contraceptive methods with their female partner from screening until 4 weeks after last dose of study drugs(except of surgical sterilization), such as complete abstinence from intercourse, condom, and their female partner use contraceptives , vaginal ring , cervical cap or contraceptive diaphragm, IUD, etc.
5. Male subjects must agree to refrain from sperm donation from the date of screening until 4 weeks after the last dose of study drugs;
6. Body mass index (BMI)≥18.0 and≤32.0 kg/m2, and Weight≥40 kg;
7. Confirmation of chronic HCV infection documented by either:

   1. A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit, or
   2. A liver biopsy performed prior to the Baseline/Day 1 visit with evidence of chronic HCV infection.
8. Serological detection of anti-HCV antibodies was positive at screening;
9. HCV RNA≥1×104 IU/mL at Screening;
10. HCV genotype 1a, 1b, or mixed 1a/1b at screening as determined by the Central Laboratory;
11. Classification as treatment naive or treatment experienced:

    1. Treatment naive is defined as having never been exposed to approved or experimental HCV-specific direct-acting antiviral agents or prior treatment of HCV with interferon (with or without ribavirin);
    2. Treatment experienced is defined as prior treatment failure to a regimen containing interferon (IFN-α,β or Peg-IFN±RBV) that was completed at least 2 months prior to screening. and the subject's medical records must include sufficient detail of prior virologic failure to allow for categorization of prior response, as either:

    i) Non-Responder: Decrease of HCV RNA<2 log at week 12 compared to baseline; ii) Partially-Responder: Decrease of HCV RNA>2 log at week 12 compared to baseline, and detectable HCV RNA levels within week 12 and week 24; iii) Breakthrough/Relapse: Subject achieved undetectable HCV RNA levels (HCV RNA < LLOQ) during treatment, but did not achieve sustained virologic response (SVR); iv) Intolerance: Subjects have discontinued interferon-based treatment due to intolerance which proved by chief complaint or medical records.
12. Absence of cirrhosis is defined as any one of the following:

    1. Liver biopsy within 2 years of Screening or at Screening showing absence of cirrhosis (e.g. Metavir score=0-3 or Ishak score<5), or
    2. Fibroscan within 6 months of Screening or at Screening with a result of ≤12.5 kPa.

    liver biopsy results will supersede fibroscan results and be considered definitive.
13. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Current or prior history of any of the following:

   1. Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage);
   2. Chronic liver disease of a non-HCV etiology (Including but not limited to hemochromatosis, Wilson's disease,alfa-1 antitrypsin deficiency);
   3. Significant cardiac disease(Including but not limited to myocardial infarction, bradycardia) ;
   4. Significant pulmonary disease;
   5. Malabsorption syndrome or gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drug;
   6. Central nervous system trauma, epilepsy, stroke or transient ischemic attack;
   7. Psychiatric illness or psychological disease or relevant medical history;
   8. Malignancy diagnosed before signing the informed consent form ( except for specific cancers that have been cured by surgical resection (basal cell skin cancer, etc) or cervical carcinoma in situ are allowed). subjects under evaluation for malignancy are not eligible;
   9. Solid organ transplantation;
   10. Subjects have any other medical disorder that may interfere with subjects treatment, assessment or compliance with the protocol.
2. Subjects has the following laboratory parameters at screening:

   1. ALT > 10×the upper limit of normal (ULN);
   2. AST > 10×ULN;
   3. Total bilirubin> 1.5 × ULN;
   4. Albumin< 3.5 g/dL;
   5. AFP>100 ng/mL; If 20 ng/mL≤AFP≤100 ng/mL, a liver ultrasound examination is required to exclude subjects suspected of hepatocellular carcinoma;
   6. INR > 1.5 x ULN;
   7. Hemoglobin<11 g/dL for female subjects; <12 g/dL for male subjects;
   8. Platelets<90 x109/L;
   9. Neutrophil absolute count< 1.5 ×109/L;
   10. HbA1c > 8.5%;
   11. Creatinine clearance (CLcr) <50 mL /min as calculated by the Cockcroft-Gault equation;
   12. HBsAg serology test results were positive;
   13. HIV antibody test results were positive.
3. Screening ECG with clinically significant abnormalities;
4. Prior exposure to approved or experimental HCV-specific direct-acting antiviral agent;
5. Use of any prohibited concomitant medications;
6. Significant drug allergy, or known hypersensitivity to DAG181, SOF and its metabolites, or formulation recipients;
7. A positive drug screen at screening will exclude subjects unless it can be explained by non-prescription drug or prescribed medication; the diagnosis and prescription must be approved by the investigator;
8. Pregnant or nursing female or male with pregnant female partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with sustained virologic response 12 weeks after discontinuation of therapy (SVR12) | Posttreatment Week 12
  SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping study treatment
Safety and tolerability were evaluated based on adverse event monitoring, laboratory tests, 12-lead ECG assessments, vital signs measurements and physical examinations. | Up to posttreatment week 24

SECONDARY OUTCOMES:
Percentage of subjects with sustained virologic response 4, 8 and 24 weeks after discontinuation of therapy (SVR4,SVR8 and SVR24) | Posttreatment Weeks 4,8 and 24
  SVR4,SVR8 and SVR24 were defined as HCV RNA < the lower limit of quantitation (LLOQ) at 4, 8 and 24 weeks after stopping study treatment, respectively.
Percentage of subjects with HCV RNA < the lower limit of quantitation (LLOQ) while on treatment | Baseline to week 12
The time to first achieve "HCV RNA < the lower limit of quantitation (LLOQ)" while on treatment | Baseline to week 12
HCV RNA change from baseline | Up to posttreatment week 24
Percentage of subjects with virologic failure | Up to posttreatment week 24
  Virologic failure was defined as:
  1. On-treatment virologic failure: Breakthrough (confirmed HCV RNA ≥the lower limit of quantitation (LLOQ) after having previously had HCV RNA <the lower limit of quantitation (LLOQ) while on treatment), or Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or Non-response (HCV RNA persistently ≥the lower limit of quantitation (LLOQ) through 8 weeks of treatment);
  2. Virologic relapse: Confirmed HCV RNA ≥the lower limit of quantitation (LLOQ) during the posttreatment period having achieved HCV RNA <the lower limit of quantitation (LLOQ) at last on-treatment visit.
Viral resistance | Up to posttreatment week 24
  Viral resistance to DAG181 and/or SOF during treatment and after cessation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, Doctor, Study Chair — Peking University People's Hospital
Locations (17):
- China (17):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University Science & Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyan Hospital, Central South University, Changsha, Hunan
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tangdu Hospital, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No